CLINICAL TRIAL: NCT06180993
Title: Evaluation of the Effectiveness and Impact of Nirsevimab Administered as Routine Immunization
Acronym: NIRSE-GAL
Status: Recruiting | Type: Observational
Sponsor: Federico Martinón Torres (Other)
Responsible Party: Sponsor-Investigator, Federico Martinón Torres, Principal investigator, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Other Study IDs: NIRSE-GAL
Record Dates: First submitted 2023-12-08; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — nirsevimab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- At birth cohort: Subjects born from September 25, 2023 to March 31 in each of the 3 RSV seasons under study 2023/2024, 2024/2025, 2025/2026
  Interventions: Biological: Nirsevimab
- Risk Cohort: Subjects with risk factors born between 1 October 2021 and 31 March 2023
  Interventions: Biological: Nirsevimab
- Catch-up cohort: Subjects born between 1 April and 24 September 2023
  Interventions: Biological: Nirsevimab

INTERVENTIONS:
Biological: Nirsevimab — Nirsevimab will be administered administered in a single dose at birth for birth cohort and at the beginning of the campaign for the other cohorts under study
  Other Names: Beyfortus

SUMMARY:
A longitudinal observational study based on routinely collected data on hospital and health care use for RSV infections will be undertaken. The Galician public health registries will be used for data collection including baseline information and follow-up data. Historical data will be retrieved for comparison purposes. The study aims to observe and analyze data from all the eligible children in Galicia for nirsevimab treatment. The number of eligible children is expected to be approximately 14,000 per each RSV season.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of nirsevimab in preventing RSV in healthy infants and high-risk children less than 24 months of age at the start of RSV season in Galicia.

The target population to receive nirsevimab is around 14,000 subjects including all healthy newborns during the RSV season, those < 6 months at the start of the season, as well as those < 24 months with comorbidities at the start of the season. Nirsevimab will be administered as part of the immunization program of Galicia and following the implementation plan designed by the Public Health authorities, using the vaccination facilities of the Galician system, i.e., hospitals and primary care centres. Appointments for administration and registration of administered doses will be performed as per usual immunization protocols. The expected coverage with nirsevimab in the target population is expected to be high (>80%).

RSV testing is routinely performed in the hospital and emergency department settings. The Galician Regional Surveillance Information System will retrieve all the existing information of the different electronic databases for new RSV cases detected in Galicia, including hospitalization, primary care, drug administration and immunization. RSV case ascertainment and classification will be per- formed by a specialized clinical team according to pre-established definitions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects born in Galicia from April 1st, 2023 and March 1st, 2026

Exclusion Criteria:

* No specific criteria has been reported

Ages: 1 Day to 24 Months | Sex: All
Age Groups: Child
Study Population: All children born between April 1st, 2023 and March 1st, 2026, both dates included, in Galicia (North- west Spain)
Sampling Method: Non-Probability Sample
Enrollment: 42000 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of RSV LRTI hospitalization through the RSV season | 8 months (from October to May)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

REFERENCES:
- [Derived] Razzini JL, Gine-Vazquez I, Jin J, Santiago-Perez MI, Perez-Martinez O, Otero-Barros MT, Suarez-Gaiche N, Kramer R, Platero-Alonso L, Alvarez-Gil RM, Ces-Ozores OM, Nartallo-Penas V, Miras-Carballal S, Pineiro-Sotelo M, Gonzalez-Perez JM, Rodriguez-Tenreiro-Sanchez C, Manzanares-Casteleiro A, Dacosta-Urbieta A, Alvarez-Smith C, Rivero-Calle I, Salas A, Duran-Parrondo C, Mallah N, Martinon-Torres F. Impact of universal nirsevimab prophylaxis in infants on hospital and primary care outcomes across two respiratory syncytial virus seasons in Galicia, Spain (NIRSE-GAL): a population-based prospective observational study. Lancet Infect Dis. 2026 Jan 12:S1473-3099(25)00742-X. doi: 10.1016/S1473-3099(25)00742-X. Online ahead of print. PMID 41539320
- [Derived] Manzanares A, Pardo-Seco J, Rivero-Calle I, Dacosta-Urbieta A, Mallah N, Santiago-Perez MI, Perez-Martinez O, Otero-Barros MT, Suarez-Gaiche N, Kramer R, Jin J, Platero-Alonso L, Alvarez-Gil RM, Ces-Ozores OM, Nartallo-Penas V, Miras-Carballal S, Pineiro-Sotelo M, Gonzalez-Perez JM, Rodriguez-Tenreiro-Sanchez C, Salas A, Duran-Parrondo C, Martinon-Torres F. Respiratory syncytial virus-related lower respiratory tract infection hospitalizations in infants receiving nirsevimab in Galicia (Spain): the NIRSE-GAL study. Eur J Pediatr. 2025 May 2;184(5):321. doi: 10.1007/s00431-025-06151-3. PMID 40314706
- [Derived] Mallah N, Ares-Gomez S, Pardo-Seco J, Malvar-Pintos A, Santiago-Perez MI, Perez-Martinez O, Otero-Barros MT, Suarez-Gaiche N, Kramer R, Jin J, Platero-Alonso L, Alvarez-Gil RM, Ces-Ozores OM, Nartallo-Penas V, Miras-Carballal S, Pineiro-Sotelo M, Gonzalez-Perez JM, Rodriguez-Tenreiro C, Rivero-Calle I, Salas A, Duran-Parrondo C, Martinon-Torres F. Assessment of effectiveness and impact of universal prophylaxis with nirsevimab for prevention of hospitalizations due to respiratory syncytial virus in infants. The NIRSE-GAL study protocol. Hum Vaccin Immunother. 2024 Dec 31;20(1):2348135. doi: 10.1080/21645515.2024.2348135. Epub 2024 May 13. PMID 38738683
- [Derived] Ares-Gomez S, Mallah N, Santiago-Perez MI, Pardo-Seco J, Perez-Martinez O, Otero-Barros MT, Suarez-Gaiche N, Kramer R, Jin J, Platero-Alonso L, Alvarez-Gil RM, Ces-Ozores OM, Nartallo-Penas V, Miras-Carballal S, Pineiro-Sotelo M, Malvar-Pintos A, Gonzalez-Perez JM, Rodriguez-Tenreiro-Sanchez C, Rivero-Calle I, Salas A, Duran-Parrondo C, Martinon-Torres F; NIRSE-GAL study group. Effectiveness and impact of universal prophylaxis with nirsevimab in infants against hospitalisation for respiratory syncytial virus in Galicia, Spain: initial results of a population-based longitudinal study. Lancet Infect Dis. 2024 Aug;24(8):817-828. doi: 10.1016/S1473-3099(24)00215-9. Epub 2024 Apr 30. PMID 38701823